CLINICAL TRIAL: NCT00982995
Title: UMCC 2008.048 Palonosetron for the Treatment of Nausea and Vomiting in Terminally Ill Patients
Brief Title: Palonosetron for the Treatment of Nausea and Vomiting in Terminally Ill Patients
Acronym: HUM21469
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: site terminated due to lack of enrollment
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UMCC 2008.048
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Nausea; Vomiting; Terminally Ill
MeSH Terms: conditions — Nausea; Vomiting | interventions — Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palonosetron (Experimental): Palonosetron 0.25 mg I.V. bolus
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Palonosetron — Palonosetron 0.25 mg as an I.V. bolus. After Palonosetron treatment, no other nausea medication will be given for 2 hours. At that point, if no relief from nausea or vomiting has occured then other anti-nausea medications may be prescribed, and patient will be taken off study. If relief from nausea and vomiting as a result of the Palonosetron occurs, patient will not receive any more anti-nausea medication unless nausea recurs. If it does recur and patient wishes to be retreated with Palonosetron. This may be repeated for a total of 3 doses, as long as it is providing relief.

SUMMARY:
The primary objective of this study is to determine the complete response (no vomiting and no need for other medications to treat nausea) in terminally ill patients suffering from nausea and/or vomiting, who are treated with palonosetron. Another objective is to determine the partial response (relief of nausea and vomiting to the extent that the patient wishes to continue treatment with palonosetron) after being treated with palonosetron. Palonosetron is currently approved by the FDA to prevent nausea and vomiting associated with chemotherapy. The investigators are testing this medication to see if it can help to relieve nausea and vomiting not associated with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years old.
2. Patient must have a terminal diagnosis, with estimated survival of 6 months or less.
3. Patients must have nausea and/or vomiting, not relieved with 1 or more anti-nausea medications. If the patient is treated with an anti-nausea medication, a minimum of 2 hours should pass to ensure that the medication is given a chance to be effective. If there is no relief after 2 hours, then the patient may be treated with palonosetron.
4. Patient's medications must be reviewed. Any medications possibly causing nausea should be stopped if possible. For example, if an opiate is suspected of causing nausea, another opiate should be substituted. However, if this is not effective, or if a medication change cannot be made, then the patient would be eligible for this study.
5. Patient must be able to understand and sign informed consent
6. Patients who have a bowel obstruction that will not be relieved by surgery may be enrolled. This includes patients whose obstruction is technically unresectable, or who are medically too ill to endure a surgery, or who refuse surgical intervention for any reason

Exclusion Criteria:

1. Patient has received chemotherapy in the past 28 days.
2. Assessment of possible causes of the nausea and vomiting should be done and recorded. If a reversible cause of the nausea is identified, that cause should be treated if possible. If the treatment relieves the nausea, then the patient is excluded from this study. Possible reversible causes of nausea and vomiting that should be excluded are:

   * Other medical conditions such as benign positional vertigo, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Urba, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palonosetron
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Palonosetron
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 65 [55 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Complete Response (no Vomiting and no Need for Nausea Rescue Medication) in Terminally Ill Patients Suffering From Nausea and/or Vomiting, Treated With Palonosetron.
Time Frame: 96 hours after dosing
Population: The study was unable to accrue the required number of patients to analyze the primary outcome.
Arm/Group | Palonosetron
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine the Partial Response (Relief of Nausea and Vomiting to the Extent That the Patient Desires Continued Dosing With Palonosetron,) in Terminally Ill Patients Suffering From Nausea and/or Vomiting, Treated With Palonosetron
Time Frame: 96 hours after dosing
Population: The study was unable to accrue the required number of patients to analyze the primary outcome.
Arm/Group | Palonosetron
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Palonosetron
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palonosetron (N=3)
Thromboembolic Event (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Accrual for the study was low. Due to issues with funding, we were unable to add a second site in order to accrue additional patients and the study was closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes